CLINICAL TRIAL: NCT01384591
Title: Pilot Study of Losartan and N-acetylcysteine as Inhibitors of Muscle Oxidative Stress in Elderly
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-091
Record Dates: First submitted 2011-06-23; First posted 2011-06-29 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Aging
Keywords: oxidative stress; blood flow; antioxidant; muscle; elderly
MeSH Terms: interventions — Acetylcysteine; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Losartan and placebo N-acetylcysteine (Experimental): losartan (25mg/dose) and placebo N-acetylcysteine (NAC) 3 total doses: 1 dose on day 1, 2 doses on day 2.
  Interventions: Drug: Losartan; Drug: Placebo N-acetylcysteine
- Placebo losartan and placebo N-acetylcysteine (Placebo Comparator): Placebo losartan and placebo N-acetylcysteine (NAC) 3 total doses: 1 dose on day 1, 2 doses on day 2.
  Interventions: Drug: Placebo losartan; Drug: Placebo N-acetylcysteine
- N-acetylcysteine and placebo losartan (Experimental): N-acetylcysteine (NAC) (50 mg/kg/dose) and placebo losartan 3 total doses: 1 dose on day 1, 2 doses on day 2.
  Interventions: Drug: N-acetylcysteine; Drug: Placebo losartan

INTERVENTIONS:
Drug: N-acetylcysteine — 50 mg/kg/dose. 3 total doses: 1 dose on day 1, 2 doses on day 2.
  Other Names: NAC
  Arms: N-acetylcysteine and placebo losartan
Drug: Losartan — 25mg/dose. 3 total doses: 1 dose on day 1, 2 doses on day 2.
  Other Names: Cozaar
  Arms: Losartan and placebo N-acetylcysteine
Drug: Placebo losartan — Placebo losartan 3 total doses: 1 dose on day 1, 2 doses on day 2.
  Other Names: Placebo
  Arms: N-acetylcysteine and placebo losartan; Placebo losartan and placebo N-acetylcysteine
Drug: Placebo N-acetylcysteine — Placebo N-acetylcysteine 3 total doses: 1 dose on day 1, 2 doses on day 2.
  Other Names: Placebo
  Arms: Losartan and placebo N-acetylcysteine; Placebo losartan and placebo N-acetylcysteine

SUMMARY:
The general hypothesis is that elderly have diminished nutritive flow to skeletal muscle and impaired capacity for building muscle. In aging populations, this decreased ability to build muscle may represent a tipping point in the progression towards chronic physical frailty and disability. The goal is to examine whether novel pharmacologic therapies can improve nutritive blood flow to the muscles and muscle building in the elderly.

The purpose of this study is 1) to determine if losartan administration will enhance blood flow and 2) to determine if N-acetylcysteine (NAC) will enhance blood flow.

The investigators will study community dwelling, healthy older men and women (60-85 years). Subjects will be randomized to one of three groups:

Experimental Group 1: Placebo losartan and placebo N-acetylcysteine (NAC). Experimental Group 2: losartan (25mg/dose) and placebo N-acetylcysteine (NAC). Experimental Group 3: N-acetylcysteine (NAC) (50 mg/kg/dose) and placebo

Subjects will admit to the clinic on day 1 of the study. Baseline testing consisting of leg blood flow (LBF), contrast enhanced ultrasound, handgrip testing and fatigue questionnaires. After testing is completed the subjects will recieve their first dose of NAC/ losartan/ placebo with dinner. Subjects will be fasted after 10 pm. On day 2, leg blood flow (LBF) will be measured approximately 12 hours post dose 1. Subjects will receive their second dose of NAC/ losartan/ placebo. Leg blood flow will be measured 1 hour and 2 hours post dose 2 of study interventions. The subjects will eat a meal and receive their third dose of the study intervention. Leg blood flow will be repeated at 1 hour and 2 hours post dose 3. Appoximately 30 minutes after dose 3 of the study intervention, handgrip testing will be performed and fatigue questionnaires completed.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 60-85 years.
2. Ability to sign informed consent.
3. Ability to sign consent form.
4. Ability to pass a mini-mental status exam (score >23 on the 30-item Mini Mental State Examination, MMSE).
5. Free-living, prior to admission.

Exclusion Criteria:

1. Subjects with cardiac abnormalities considered exclusionary by the study physicians (e.g., unstable angina or a cardiology-confirmed ECG that demonstrates cardiac abnormalities such as > 0.2 mV horizontal or downsloping ST segment depression, frequent arrhythmia's (> 10 PVC/min), or valvular disease).
2. Subjects with uncontrolled metabolic disease, including liver or renal disease.
3. Subjects with vascular disease characterized by a combination of risk factors of peripheral atherosclerosis. (e.g., uncontrolled hypertension, obesity, uncontrolled diabetes, hypercholesterolemia > 250 mg/dl, claudication or evidence of venous or arterial insufficiency upon palpitation of femoral, popliteal, and pedal arteries.
4. Any history of hypo- or hyper-coagulation disorders. (e.g., Coumadin use or history of DVT or PE).
5. Subjects with chronically elevated systolic pressure >170 or a diastolic blood pressure > 100. Subjects may be included if they are taking medication and have a blood pressure below these criteria.
6. Subjects with cancer or recently (6 months) treated cancer other than basal cell carcinoma.
7. Any subject currently on a weight-loss diet or a body mass index > 33 kg/m2.
8. Inability to abstain from smoking for duration of study.
9. A history of > 20 pack per year smoking.
10. Subjects with atrial fibrillation, history of syncope, angina, or congestive heart failure.
11. Any subject that is HIV-seropositive or has active hepatitis.
12. Recent anabolic or corticosteroids use (within 3 months).
13. Subjects with low hemoglobin or hematocrit (i.e., lower than accepted lab values).
14. Agitation/aggression disorder.
15. Dementia.
16. History of stroke with motor disability.
17. A recent history (<12 months) of GI bleed.
18. Alcohol (more than 3 drinks per day) or drug abuse.
19. Polycystic ovary syndrome (PCOS) and/or hyperthecosis.
20. Non-classical adrenal hyperplasia.
21. Cushing's syndrome.
22. Pregnancy.
23. Hyperprolactinoma, hypothyroidism.
24. Lactose intolerance.
25. Subjects with coronary heart or mitral valvular rheumatic heart disease.
26. Subjects with impaired renal function and/or renal artery stenosis.
27. Subjects with pulmonary hypertension.
28. Subjects on any medications known to vasodilate the peripheral arteries.
29. Subjects taking NSAIDs
30. Physical dependence or frailty (impairment of activities of daily living, ADLs).
31. History of falls (>2/year).
32. Depression (>5 of the 15 items on the Geriatric Depression Scale (GDS).
33. Subjects suffering malnutrition or with a BMI < 20 kg/m2 with low albumin or transferrin.
34. Asthma
35. Any other condition or event considered exclusionary by the PI and covering faculty physician.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — UTMB; Astrid M Horstman, PhD, Study Director — UTMB
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Losartan and Placebo N-acetylcysteine | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan and Placebo N-acetylcysteine | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 2 | 2 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (3.6) | 72.3 (2.1) | 68.5 (1.3) | 72 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 1 | 2 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 2 | 6
Total Mass [Mean (Standard Deviation); unit: kilograms] | 67.1 (10.2) | 72.7 (11.4) | 65.7 (3.5) | 68.5 (7.8)
Lean Body Mass [Mean (Standard Deviation); unit: kilograms] | 41.2 (11.1) | 52.9 (14.2) | 45.9 (2.4) | 46.7 (9.7)
Fat Mass [Mean (Standard Deviation); unit: kilograms] | 23.7 (0.98) | 16.6 (3.2) | 16.8 (0.490) | 19.1 (3.90)

OUTCOME MEASURES:

1. Primary Outcome: Leg Blood Flow as Measured by Doppler Ultrasound
Description: Femoral Doppler Blood Flow was evaluated via Doppler ultrasound. For the two-dimensional (2-D) and Doppler ultrasound measurements, an ultrasound system (HDI-5000; Philips Medical Systems, Bothell, WA) with a linear array transducer (L7-4) was used with a transmit frequency of 12MHz. 2-D imaging of the common femoral artery will be performed in the long axis. Images will be triggered to the R wave of the cardiac cycle, and the femoral artery diameter will be measured using online video calipers. A pulsed-wave Doppler sample blood volume will be placed at the same location in the center of the artery, and the mean blood velocity will be measured using online angle correction and analysis software. Femoral artery mean blood flow will be calculated from 2-D and Doppler ultrasound data using the equation: Q = vπ ∙ (d/2)2, where Q is femoral blood flow, v is mean femoral artery blood flow velocity, and d is femoral artery diameter.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
ml/minute | 174.99 (176.02) | 102.08 (3.42) | 428.45 (114.57)

2. Primary Outcome: Leg Blood Flow as Measured by Doppler Ultrasound
Description: as for outcome 1
Time Frame: 12 hours post dose one of the intervention
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
ml/minute | 181.88 (204.92) | 69.83 (77.57) | 91.68 (4.88)

3. Primary Outcome: Leg Blood Flow as Measured by Doppler Ultrasound
Description: as for outcome 1
Time Frame: 1 hour post dose two of the intervention, average of 13 hours post dose 1 of the intervention
Population: Missed blood flow measurement on one placebo participant at this time point.
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 1 | 2 | 2
ml/minute | 105.80 | 90.06 (39.19) | 95.60 (64.67)

4. Primary Outcome: Leg Blood Flow as Measured by Doppler Ultrasound
Description: as for outcome 1
Time Frame: 2 hours post dose two of the intervention, average of 14 hours post dose one of the intervention
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
ml/minute | 214.56 (88.42) | 70.37 (15.35) | 114.34 (38.71)

5. Primary Outcome: Leg Blood Flow as Measured by Doppler Ultrasound
Description: as for outcome 1
Time Frame: Post dose three of the intervention and a meal, average of 17 hours post dose one of the intervention
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
ml/minute | 158.71 (83.85) | 109.94 (59.51) | 153.38 (103.37)

6. Primary Outcome: Leg Blood Flow as Measured by Doppler Ultrasound
Description: as for outcome 1
Time Frame: 1 hour post dose three of the intervention and a meal, average of 18 hours post dose one of the intervention
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
ml/minute | 84.41 (18.57) | 104.40 (56.55) | 152.10 (46.59)

7. Primary Outcome: Leg Blood Flow as Measured by Doppler Ultrasound
Description: as for outcome 1
Time Frame: 2 hours post dose three of the intervention and a meal, average of 19 hours post dose one of the intervention
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
ml/minute | 70.60 (17.46) | 128.78 (123.74) | 57.79 (29.24)

8. Secondary Outcome: Handgrip Strength of Dominant Hand as Measured by Handgrip Dynamometry at 50% Perceived Effort at Baseline
Description: Handgrip Strength of dominant hand is measured by handgrip dynamometry at 50% perceived effort with subjects performing one set of three contractions.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
kilograms | 21.5 (6.5) | 23.2 (4.9) | 20.5 (16.7)

9. Secondary Outcome: Handgrip Strength of Non-dominant Hand as Measured by Handgrip Dynamometry at 50% Perceived Effort at Baseline
Description: Handgrip Strength of non-dominant hand is measured by handgrip dynamometry at 50% perceived effort with subjects performing one set of three contractions.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
kilograms | 24.2 (2.6) | 19.3 (1.9) | 17.0 (15.1)

10. Secondary Outcome: Handgrip Strength of Dominant Hand as Measured by Handgrip Dynamometry at 100% Effort at Baseline
Description: Handgrip Strength of dominant hand is measured by handgrip dynamometry at 100% effort with subjects performing one set of three contractions.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
kilograms | 45.2 (8.2) | 33.2 (4.0) | 28.8 (13.9)

11. Secondary Outcome: Handgrip Strength of Non-dominant Hand as Measured by Handgrip Dynamometry at 100% Effort at Baseline
Description: Handgrip Strength of non-dominant hand is measured by handgrip dynamometry at 100% effort with subjects performing one set of three contractions.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
kilograms | 47.1 (7.9) | 31.1 (0.8) | 26.5 (11.1)

12. Secondary Outcome: Handgrip Fatigue of Dominant Hand as Measured by Handgrip Dynamometry at Baseline
Description: Handgrip fatigue of dominant hand as measured by handgrip dynamometry fatigue test. The non-dominant hand hold a continuous contraction at 20% of the subjects maximal voluntary contraction for 5 minutes. Data is reported as % of Maximal Voluntary Contraction after fatigue test.
Time Frame: baseline
Population: Data for 2 subjects wasn't recorded.
Measure: Mean (Standard Deviation); unit: % of Maximal Voluntary Contraction
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 1 | 2 | 1
% of Maximal Voluntary Contraction | 129.6 | 94.2 (12.06) | 103.4

13. Secondary Outcome: Handgrip Fatigue of Non-dominant Hand as Measured by Handgrip Dynamometry at Baseline
Description: Handgrip fatigue of non-dominant hand as measured by handgrip dynamometry fatigue test. The non-dominant hand hold a continuous contraction at 20% of the subjects maximal voluntary contraction for 5 minutes. Data is reported as % of Maximal Voluntary Contraction (MVC) after fatigue test.
Time Frame: baseline
Population: Data for 2 subjects was not recorded.
Measure: Mean (Standard Deviation); unit: % of Maximal Voluntary Contraction
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 1 | 2 | 1
% of Maximal Voluntary Contraction | 64.55 | 83.62 (2.33) | 90.29

14. Secondary Outcome: Handgrip Strength of Dominant Hand as Measured by Handgrip Dynamometry at 50% Perceived Effort After All Doses of Study Intervention
Description: as for outcome 8
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
kilograms | 21.2 (13.9) | 15.8 (1.6) | 16.2 (11.1)

15. Secondary Outcome: Handgrip Strength of Non-dominant Hand as Measured by Handgrip Dynamometry at 50% Perceived Effort After All Doses of Study Intervention
Description: as for outcome 9
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
kilograms | 17.8 (4.5) | 14.8 (4.5) | 13.7 (7.1)

16. Secondary Outcome: Handgrip Strength of Dominant Hand as Measured by Handgrip Dynamometry at 100% Perceived Effort After All Doses of Study Intervention
Description: Handgrip Strength of dominant hand is measured by handgrip dynamometry at 100% perceived effort with subjects performing one set of three contractions.
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
kilograms | 44.1 (6.2) | 31.3 (6.6) | 24.2 (13.0)

17. Secondary Outcome: Handgrip Strength of Non-dominant Hand as Measured by Handgrip Dynamometry at 100% Perceived Effort After All Doses of Study Intervention
Description: Handgrip Strength of non-dominant hand is measured by handgrip dynamometry at 100% perceived effort with subjects performing one set of three contractions.
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
kilograms | 42.3 (3.9) | 28.6 (2.7) | 30.2 (0.2)

18. Secondary Outcome: Handgrip Fatigue of Dominant Hand as Measured by Handgrip Dynamometry After All Doses of Study Intervention
Description: Handgrip fatigue of dominant hand as measured by handgrip dynamometry fatigue test. The non-dominant hand hold a continuous contraction at 20% of the subjects maximal voluntary contraction for 5 minutes. Data reported as % of Maximal Voluntary Contraction (MVC) after fatigue test.
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Population: Data for 2 subjects not recorded.
Measure: Mean (Standard Deviation); unit: % of Maximal Voluntary Contraction
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 1 | 2 | 1
% of Maximal Voluntary Contraction | 101.0 | 95.97 (2.16) | 111

19. Secondary Outcome: Handgrip Fatigue of Non-dominant Hand as Measured by Handgrip Dynamometry After All Doses of Study Intervention
Description: Handgrip fatigue of non-dominant hand as measured by handgrip dynamometry fatigue test. The non-dominant hand hold a continuous contraction at 20% of the subjects maximal voluntary contraction for 5 minutes. Data reported as % of Maximal Voluntary Contraction (MVC) after fatigue test.
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Population: Data from 2 subjects was not recorded.
Measure: Mean (Standard Deviation); unit: % of Maximal Voluntary Contraction
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 1 | 2 | 1
% of Maximal Voluntary Contraction | 88.61 | 93.25 (11.32) | 95.60

20. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale General Fatigue at Baseline
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the general fatigue scale is 24 to 0, with the higher number meaning more fatigue.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0 (0) | 1.5 (2.12) | 3.5 (2.11)

21. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale General Fatigue After All Doses of Study Intervention
Description: as for outcome 20
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0 (0) | 2 (2.8) | 6.5 (0.7)

22. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale Physical Fatigue at Baseline
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the physical fatigue scale is 24 to 0, with the higher number meaning more fatigue.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0.5 (0.7) | 0.5 (0.7) | 3 (1.4)

23. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale Physical Fatigue After All Doses of Study Intervention
Description: as for outcome 22
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0 (0) | 0.5 (0.7) | 7 (1.4)

24. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale Emotional Fatigue at Baseline
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the emotional fatigue scale is 24 to 0, with the higher number meaning more fatigue.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0.5 (0.7) | 0 (0) | 4 (5.6)

25. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale Emotional Fatigue After All Doses of Study Intervention
Description: as for outcome 24
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0.5 (0.7) | 0 (0) | 7.5 (2.12)

26. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale Mental Fatigue at Baseline
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the mental fatigue scale is 24 to 0, with the higher number meaning more fatigue.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0.5 (0.7) | 0.5 (0.7) | 4.5 (0.7)

27. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale Mental Fatigue After All Doses of Study Intervention
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the mental fatigue scale is 24 to 0, with the higher number meaning more fatigue
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0 (0) | 1 (1.4) | 6.5 (0.7)

28. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale Vigor Fatigue at Baseline
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the vigor scale is 0 to 24, with the higher number meaning more vigor.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 18 (0) | 15 (2.8) | 16.5 (3.5)

29. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Subscale Vigor Fatigue After All Doses of Study Intervention
Description: as for outcome 28
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 20.5 (3.5) | 15.5 (3.5) | 14 (1.4)

30. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Total Score at Baseline
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | -16.5 (2.12) | -12.5 (6.36) | -1.5 (4.95)

31. Secondary Outcome: Personal Perceptual Fatigue Measured by Multidimensional Fatigue Symptom Inventory - Total Score After All Doses of Study Intervention
Description: as for outcome 30
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | -20 (2.8) | -12 (1.4) | 13.5 (2.12)

32. Secondary Outcome: Global Fatigue Score as Measured by Brief Fatigue Inventory at Baseline
Description: The Brief Fatigue Inventory is a 9 item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life), with "0" being no fatigue and "10" being as bad as you can imagine. The Global Fatigue score is calculated by averaging the answers of all the questions. Score ranges (0 to 10) with higher score indicating a worse outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0.55 (0.78) | 0.38 (0.39) | 1.11 (0.16)

33. Secondary Outcome: Global Fatigue Score as Measured by Brief Fatigue Inventory After Study Invention
Description: The Brief Fatigue Inventory is a 9 item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life), with "0" being no fatigue and "10" being as bad as you can imagine. The Global Fatigue score is calculated by averaging the answers of all the questions. Score range 0 to 10, with a higher score indicating a worse outcome.
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0.5 (0.7) | 0.22 (0.31) | 1.19 (0.43)

34. Secondary Outcome: Perceptual Fatigue of Non-dominant Arm as Measured by Visual Analog Scale Before Handgrip Fatigue Test at Baseline.
Description: The Visual Analog Scale for Fatigue is an 11cm long line. The subject is asked to mark their level of fatigue (0cm being no fatigue and 11cm being extreme fatigue). This test was performed before and after the handgrip fatigue test, where the non-dominant hand hold a continuous contraction at 20% of the subjects maximal voluntary contraction for 5 minutes.
  Handgrip testing was performed at baseline (before any intervention) and post dose three of the intervention, average of 17 hours post dose one intervention.
Time Frame: baseline - before handgrip fatigue test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0.3 (0.14) | 3.3 (2.69) | 0.2 (0.28)

35. Secondary Outcome: Perceptual Fatigue of Non-dominant Arm as Measured by Visual Analog Scale After Handgrip Fatigue Test at Baseline.
Description: as for outcome 34
Time Frame: baseline - directly after handgrip fatigue test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 2.7 (3.39) | 7.5 (4.5) | 0.6 (0.84)

36. Secondary Outcome: Perceptual Fatigue of Non-dominant Arm as Measured by Visual Analog Scale Before Handgrip Fatigue Test After Study Intervention
Description: as for outcome 34
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention - Before handgrip fatigue test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 1.45 (1.62) | 1 (1.41) | 0.65 (0.92)

37. Secondary Outcome: Perceptual Fatigue of Non-dominant Arm as Measured by Visual Analog Scale After Handgrip Fatigue Test After Study Intervention
Description: as for outcome 34
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention - Directly after handgrip fatigue test
Population: Data for 1 subject was not collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 1 | 2
units on a scale | 3.4 (4.38) | 11 | 0.75 (1.06)

38. Secondary Outcome: Perceptual Fatigue of Whole Body as Measured by Visual Analog Scale Before Handgrip Fatigue Test at Baseline.
Description: as for outcome 34
Time Frame: baseline - before handgrip fatigue test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0.4 (0.14) | 1.15 (0.35) | 0.55 (0.77)

39. Secondary Outcome: Perceptual Fatigue of Whole Body as Measured by Visual Analog Scale After Handgrip Fatigue Test at Baseline.
Description: as for outcome 34
Time Frame: baseline - directly after handgrip fatigue test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 1.05 (1.20) | 5 (3.11) | 0.6 (0.85)

40. Secondary Outcome: Perceptual Fatigue of Whole Body as Measured by Visual Analog Scale Before Handgrip Fatigue Test After Study Intervention
Description: as for outcome 34
Time Frame: Post dose three of the intervention, average of 17 hours post dose one intervention - Before handgrip fatigue test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 2 | 2
units on a scale | 0.7 (0.42) | 4.1 (4.1) | 0.55 (0.77)

41. Secondary Outcome: Perceptual Fatigue of Whole Body as Measured by Visual Analog Scale After Handgrip Fatigue Test After Study Intervention
Description: as for outcome 34
Time Frame: as for outcome 37
Population: Data for 1 subject was not recorded
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
Number analyzed (Participants) | 2 | 1 | 2
units on a scale | 1.25 (1.34) | 5.3 | 0.95 (1.34)

ADVERSE EVENTS:
Arm/Group | Placebo Losartan and Placebo N-acetylcysteine | N-acetylcysteine and Placebo Losartan | Losartan and Placebo N-acetylcysteine
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Losartan and Placebo N-acetylcysteine (N=2) | N-acetylcysteine and Placebo Losartan (N=2) | Losartan and Placebo N-acetylcysteine (N=2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Rash after infusion with Definity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No